CLINICAL TRIAL: NCT02743221
Title: An Open-label, Randomised, Non-comparative Phase 2 Study Evaluating S 95005 (TAS-102) Plus Bevacizumab and Capecitabine Plus Bevacizumab in Patients With Previously Untreated Metastatic COlorectal Cancer Who Are Non-eligible for Intensive Therapy (TASCO1 Study).
Brief Title: A Study Evaluating S 95005 Plus Bevacizumab and Capecitabine Plus Bevacizumab in Patients With Previously Untreated Colorectal Cancer Who Are Non-eligible for Intensive Therapy
Acronym: TASCO1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut de Recherches Internationales Servier (Other)
Collaborators: ADIR, a Servier Group company (Industry)
Responsible Party: Sponsor
Organization: Servier (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CL2-95005-002; 2015-004544-18 (EudraCT Number)
Record Dates: First submitted 2016-02-24; First posted 2016-04-19 (Estimated); Results first posted 2019-04-16 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-07

CONDITIONS: Metastatic Colorectal Cancer
Keywords: metastatic; colorectal; cancer; untreated; first-line; S95005 (Trifluridine/tipiracil); bevacizumab; capecitabine
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Neoplasms | interventions — Trifluridine; tipiracil; Bevacizumab; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Trifluridine/tipiracil + bevacizumab (Experimental): Trifluridine/tipiracil (S95005): film-coated tablets containing 15mg of trifluridine and 7.065mg of tipiracil hydrochloride, or 20mg of trifluridine and 9.42mg of tipiracil hydrochloride.
  Bevacizumab: concentrate for solution for IV infusion containing 25mg/ml of bevacizumab.
  Trifluridine/tipiracil was administered at 35 mg/m2/dose orally within 1 hour after completion of morning and evening meals, for 5 days on/2 days off, over 2 weeks, followed by a 14-day rest period, with bevacizumab administered intravenously at the dose of 5 mg/kg every 2 weeks at Day 1 and Day 15.This treatment cycle was repeated every 4 weeks.
  Interventions: Drug: Trifluridine/tipiracil + bevacizumab
- Capecitabine + bevacizumab (Active Comparator): Capecitabine was administered at 1250 mg/m² orally BID (bis in die)on Days 1-14 of each cycle, with bevacizumab (7.5 mg/kg, IV) administered on Day 1 of each cycle. This treatment cycle was repeated every 3 weeks
  Interventions: Drug: Capecitabine + bevacizumab

INTERVENTIONS:
Drug: Trifluridine/tipiracil + bevacizumab — Patients were treated withTrifluridine/tipiracil + bevacizumab regimen until they met a discontinuation criterion.
  Arms: Trifluridine/tipiracil + bevacizumab
Drug: Capecitabine + bevacizumab — Patients were treated with capecitabine+ bevacizumab regimen until they met a discontinuation criterion.
  Arms: Capecitabine + bevacizumab

SUMMARY:
The main purpose of this study is to evaluate the progression-free survival (PFS) in patients receiving S 95005 + bevacizumab (experimental arm) or capecitabine + bevacizumab (control arm) as first-line treatment for unresectable metastatic colorectal cancer in patients non-eligible for intensive therapy.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained.
* Has ECOG (Eastern Cooperative Oncology Group) performance status of 0, 1 or 2 at the time of the randomisation.
* Has definitive histologically or cytologically confirmed adenocarcinoma of the colon or rectum.
* RAS status must have been determined (mutant or wild).
* Has at least one measurable metastatic lesion.
* No previous systemic anticancer therapy for unresectable metastatic colorectal cancer.
* Previous adjuvant (or neoadjuvant for patients with rectal cancer) chemotherapy is allowed only if if it has been completed more than 6 months before start of study treatment.
* Patient is not a candidate for combination chemotherapy with irinotecan or oxaliplatin, or for curative resection of metastatic lesions.
* Is able to take medication orally (i.e., no feeding tube).
* Has adequate organ function.
* Coagulation parameters in normal limit (or in therapeutic limit for patients treated with anticoagulant drugs).
* Women of childbearing potential must have been tested negative in a serum pregnancy test. Female participants of childbearing potential and male participants with partners of childbearing potential must agree to use a highly effective method of birth control. Women and female partners using hormonal contraceptive must also use a barrier method.

Exclusion Criteria:

* Is a pregnant or lactating female.
* Has certain serious illness or serious medical condition(s) as described in the protocol.
* Has had certain other recent treatment e.g. major surgery, field radiation, received investigational agent, within the specified time frames prior to randomisation.
* Has previously received Trifluridine/tipiracil or history of allergic reactions attributed to compounds of similar composition to Trifluridine/tipiracil or any of its excipients.
* Has rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption.
* Has contra-indication to bevacizumab or capecitabine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2016-04-29 (Actual); Primary Completion 2018-01-15 (Actual); Study Completion 2020-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Van Custem, Prof, Principal Investigator — Leuven Cancer Institute, University Hospitals Leuven
Locations (57):
- Australia (4):
  - Chris O'Brien Lifehouse Oncology, Camperdown
  - Austin Hospital Olivia Newton-John Cancer & Wellness Centre, Heidelberg
  - Western Health, Sunshine Hospital, Saint Albans
  - The Queen Elizabeth Hospital Haematology and Oncology Unit, Woodville
- Belgium (3):
  - Grand Hôpital de Charleroi Oncologie-Hématologie, Charleroi
  - UZ Leuven Campus Gasthuisberg Digestieve Oncologie, Leuven
  - CHC Saint-Joseph Oncologie-Hématoimmunopathologie, Liège
- Brazil (5):
  - Hospital do Câncer de Barretos - Fundação Pio XII, Barretos
  - Centro de Pesquisa Hospital de Caridade de Ijuí, Ijuí
  - Instituto Nacional do Câncer - INCA Unidade de Pesquisa ClínicaInstituto Nacional do Câncer - INCA Unidade de Pesquisa Clínica, Rio de Janeiro
  - Hospital de Base, Centro Intergrado de Pesquisa, São José do Rio Preto
  - Instituto do Câncer do Estado de São Paulo - ICESP, Núcleo de Pesquisa, São Paulo
- Denmark (2):
  - Rigshospitalet - Dpt of Oncology, Copenhagen
  - Odense Universitetshospital - Department of Oncology, Odense
- France (3):
  - CHU Jean Minjoz, Service d'oncologie médicale, Besançon
  - Hôpital Saint Antoine, oncology department, Paris
  - Centre René Gauducheau, Oncologie Médicale, Saint-Herblain
- Germany (3):
  - Onkologische Schwerpunktpraxis Kurfürstendamm, Berlin
  - Schwerpunktpraxis für Hämatologie und Onkologie, Magdeburg
  - Städtisches Krankenhaus München Neuperlach, Klinik für Onkologie und Hämatologie, Munich
- Italy (5):
  - Fondazione Poliambulanza Istituto Ospedaliero, Clinical Oncology, Brescia
  - A.O.U. SanMartino-IST, Unità Operativa Oncologia Medica 1, Genova
  - A.O. Ospedale Niguarda Ca' Granda-Milano, Department of Onco-Haematology- Onoclogia Falck, Milan
  - Seconda Università degli Studi di Napoli, U.O.C. di Oncologia Medica ed Ematologia, Naples
  - .O.U. Pisana-Ospedale Santa Chiara, U.O. di Oncologia Medica 2, Pisa
- Netherlands (9):
  - AMC Academisch Medisch Centrum Medische Oncologie, Amsterdam
  - Amphia Ziekenhuis, Interne Geneeskunde/Oncologie, Langendijk 75, Breda
  - Catharina Ziekenhuis, Interne Geneeskunde/Oncologie, Eindhoven
  - Martini Ziekenhuizen, Interne Geneeskunde/Oncologie, Van Swietenplein 1, Groningen
  - Tergooi Hilversum, Medische Oncologie, Van Riebeeckweg 212, Hilversum
  - Zuyderland Medisch Centrum Interne Geneeskunde, Sittard
  - Sint Antonius Ziekenhuis Interne Geneeskunde/Oncologie, Utrecht
  - VieCurie Medisch Centrum, Interne Geneeskunde, Tegelseweg 210, Venlo
  - Isala Klinieken, Medische oncologie, Dokter Van Heeweg 2, Zwolle
- Poland (4):
  - Szpitale Pomorskie Sp. z o.o. Oddzial Onkologii i Radioterapii, Gdynia
  - SP ZOZ Szpital Uniwersytecki w Krakowie Oddzial Kliniczny Onkologii, Krakow
  - Centralny Szpital Kliniczny MSW Klinika Onkologii i Hematologii, Warsaw
  - NZOZ MAGODENT Oddzial Onkologii Klinicznej / Chemioterapii, Warsaw
- Russia (4):
  - Russian Cancer Research Center n.a. NN Blokhin, Moscow
  - Moscow City Oncology Hospital # 62, Chemotherapy, Moscow
  - Russian Cancer Research Center n.a. NN Blokhin, Department of Research for New Antitumour Medicines, Moscow
  - Scientific Centre for Specialized Medical Care (oncological), Saint Petersburg
- Spain (8):
  - Hospital Valle de Hebrón, Servicio de Oncología, Barcelona
  - Hospital Universitario Reina Sofia, Deparatmento Oncología Médica, Córdoba
  - Instituto Catalan De Oncología, Hospitalet de Llobregat, L'Hospitalet de Llobregat
  - Hospital Universitario Gregorio Maranon, Madrid
  - Hospital Ramón y Cajal, Oncología Médica, Madrid
  - H. Universitario La Paz Oncología Médica, Madrid
  - Hospital General Universitario, Oncología Médica, Málaga
  - Complejo Hospitalario de Navarra, Oncología Médica, Pamplona
- United Kingdom (7):
  - The Beatson West of Scotland Cancer Centre GI cancers, Glasgow
  - Leicester Royal Infirmary, The HOPE Clinical Trials Unit, Leicester
  - Hammersmith Hospital, London
  - Imperial healthcare NHS Trust Charing Cross Hospital, London
  - Christie Hospital NHS Foundation Trust, GI & Endocrine, Manchester
  - Mount Vernon Hospital Department of Oncology, Northwood
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Qualified scientific and medical researchers can request access to anonymized patient-level and study-level clinical trial data.
  Access can be requested for all interventional clinical studies:
  * used for Marketing Authorization (MA) of medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * where Servier is the Marketing Authorization Holder (MAH). The date of the first MA of the new medicine (or the new indication) in one of the EEA Member States will be considered for this scope.
  In addition, access can be requested for all interventional clinical studies in patients:
  * sponsored by Servier
  * with a first patient enrolled as of 1 January 2004 onwards
  * for New Chemical Entity or New Biological Entity (new pharmaceutical form excluded) for which development has been terminated before any Marketing authorization (MA) approval.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorisation in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.
URL: http://clinicaltrials.servier.com

REFERENCES:
- [Background] Van Cutsem E, Danielewicz I, Saunders MP, Pfeiffer P, Argiles G, Borg C, Glynne-Jones R, Punt CJA, Van de Wouw AJ, Fedyanin M, Stroyakovskiy D, Kroening H, Garcia-Alfonso P, Wasan H, Falcone A, Fougeray R, Egorov A, Amellal N, Moiseyenko V. First-line trifluridine/tipiracil + bevacizumab in patients with unresectable metastatic colorectal cancer: final survival analysis in the TASCO1 study. Br J Cancer. 2022 Jun;126(11):1548-1554. doi: 10.1038/s41416-022-01737-2. Epub 2022 Apr 19. PMID 35440667
- [Derived] Van Cutsem E, Danielewicz I, Saunders MP, Pfeiffer P, Argiles G, Borg C, Glynne-Jones R, Punt CJA, Van de Wouw AJ, Fedyanin M, Stroyakovskiy D, Kroening H, Garcia-Alfonso P, Wasan H, Falcone A, Kanehisa A, Egorov A, Aubel P, Amellal N, Moiseenko V. Trifluridine/tipiracil plus bevacizumab in patients with untreated metastatic colorectal cancer ineligible for intensive therapy: the randomized TASCO1 study. Ann Oncol. 2020 Sep;31(9):1160-1168. doi: 10.1016/j.annonc.2020.05.024. Epub 2020 Jun 1. PMID 32497736
- Available data/document: Individual Participant Data Set — http://clinicaltrials.servier.com/
- Available data/document: Study Protocol — https://clinicaltrials.servier.com/
- Available data/document: Statistical Analysis Plan — https://clinicaltrials.servier.com/
- Available data/document: Informed Consent Form — https://clinicaltrials.servier.com/
- Available data/document: Clinical Study Report — https://clinicaltrials.servier.com/
- Available data/document: study-level clinical trial data — https://clinicaltrials.servier.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 154 patients were randomized among whom one was deemed ineligible after randomization.
Groups:
- Trifluridine/Tipiracil + Bevacizumab: Trifluridine/tipiracil (S95005): film-coated tablets containing 15mg of trifluridine and 7.065mg of tipiracil hydrochloride, or 20mg of trifluridine and 9.42mg of tipiracil hydrochloride.
  Bevacizumab: concentrate for solution for IV infusion containing 25mg/ml of bevacizumab.
  Trifluridine/tipiracil was administered at 35 mg/m2/dose orally within 1 hour after completion of morning and evening meals, for 5 days on/2 days off, over 2 weeks, followed by a 14-day rest period, with bevacizumab administered intravenously at the dose of 5 mg/kg every 2 weeks at Day 1 and Day 15.This treatment cycle was repeated every 4 weeks.
  Trifluridine/tipiracil + bevacizumab: Patients were treated withTrifluridine/tipiracil + bevacizumab regimen until they met a discontinuation criterion.
- Capecitabine + Bevacizumab: Capecitabine was administered at 1250 mg/m² orally BID on Days 1-14 of each cycle, with bevacizumab (7.5 mg/kg, IV) administered on Day 1 of each cycle. This treatment cycle was repeated every 3 weeks
  Capecitabine + bevacizumab: Patients were treated with capecitabine+ bevacizumab regimen until they met a discontinuation criterion.
Period: Overall Study
Arm/Group | Trifluridine/Tipiracil + Bevacizumab | Capecitabine + Bevacizumab
Started | 77 | 77
Completed (Of note, these patients were still under treatment at the primary completion date (cut-off date).) | 21 | 17
Not Completed | 56 | 60
Not completed — Progressive disease | 29 | 38
Not completed — Adverse Event | 17 | 14
Not completed — non medical reason | 8 | 2
Not completed — Physician Decision | 2 | 5
Not completed — Patient not eligible, not treated | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Trifluridine/Tipiracil + Bevacizumab | Capecitabine + Bevacizumab | Total
Number analyzed (Participants) | 77 | 77 | 154
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 16 | 36
  >=65 years | 57 | 61 | 118
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.8 (10.2) | 72.8 (11.0) | 71.3 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 29 | 66
  Male | 40 | 48 | 88
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 73 | 72 | 145
  Asian | 1 | 2 | 3
  Other | 1 | 1 | 2
  Not collected | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: The progression free survival (PFS), defined as the time from the date of randomisation until the date of the investigator-assessed radiological disease progression or death due to any cause according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. Progressive disease (PD) was defined at least a 20% increase in the sum of diameters of target lesions (taking as reference the smallest sum on study) and an absolute increase of at least 5 mm in the sum of lesions or the appearance of new lesions.
Time Frame: Baseline and every 8 weeks (maximum follow-up duration: 17.9 months)
Population: Full Analysis Set (FAS): all randomised patients who have taken at least one dose of study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trifluridine/Tipiracil + Bevacizumab | Capecitabine + Bevacizumab
Number analyzed (Participants) | 77 | 76
months | 9.2 [7.6 to 11.6] | 7.8 [5.5 to 10.2]
Statistical Analysis 1: Comparison: Trifluridine/Tipiracil + Bevacizumab vs Capecitabine + Bevacizumab; Test type: Other — This was a non-comparative study; p = 0.09, Cox proportional hazard model; Cox proportional hazard model with adjustment for the stratification factors (RAS status, performance status ECOG); Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.48 to 1.06]

2. Secondary Outcome: Overall Response Rate (ORR)
Description: As per RECIST v1.1, Complete Response (CR) was disappearance of all target lesions; Partial Response (PR) was at least 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. The ORR was the proportion of patients who presented CR or PR with confirmation at subsequent time point or at least 4 weeks later.
Time Frame: Baseline and every 8 weeks (maximum follow-up duration: 17.9 months)
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Trifluridine/Tipiracil + Bevacizumab | Capecitabine + Bevacizumab
Number analyzed (Participants) | 77 | 76
Participants | 26 | 23
Statistical Analysis 1: Comparison: Trifluridine/Tipiracil + Bevacizumab vs Capecitabine + Bevacizumab; Test type: Other; p = 0.73, Fisher Exact

3. Secondary Outcome: Duration of Response (DR)
Description: The DR was calculated among patients with CR or PR as the time (months) from the first documentation of response to the first documentation of objective tumor progression or death due to any cause, whichever occurred first.
Time Frame: Baseline and every 8 weeks (maximum follow-up duration: 16.6 months)
Population: Tumour Response population: patients with measurable disease at baseline and with at least one tumour evaluation while on treatment.
Measure: Median (80% Confidence Interval); unit: months
Arm/Group | Trifluridine/Tipiracil + Bevacizumab | Capecitabine + Bevacizumab
Number analyzed (Participants) | 74 | 73
months | 7.9 [6.01 to 14.75] | 9.9 [8.41 to 10.02]
Statistical Analysis 1: Comparison: Trifluridine/Tipiracil + Bevacizumab vs Capecitabine + Bevacizumab; Test type: Other; Hazard Ratio (HR) = 1.16, 95% CI 2-sided [0.49 to 2.74]

4. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR was the proportion of patients with confirmed CR, PR or stable disease (SD) as best overall response. SD defined as neither sufficient decrease to qualify for PR nor sufficient increase to qualify for PD.
Time Frame: Baseline and every 8 weeks (maximum follow-up duration: 17.9 months)
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Trifluridine/Tipiracil + Bevacizumab | Capecitabine + Bevacizumab
Number analyzed (Participants) | 77 | 76
Participants | 66 | 59
Statistical Analysis 1: Comparison: Trifluridine/Tipiracil + Bevacizumab vs Capecitabine + Bevacizumab; Test type: Other; p = 0.22, Fisher Exact

5. Secondary Outcome: Overall Survival (OS)
Description: The OS was defined as the time from the date of randomisation to the date of death. If death was not confirmed, or patient was alive at study cut-off date, survival time was censored at the date of last follow-up or at the study cut-off date, whichever was earlier.
Time Frame: Baseline up to death or study cut-off (maximum follow-up duration: 19.9 months)
Population: FAS
Measure: Median (80% Confidence Interval); unit: months
Arm/Group | Trifluridine/Tipiracil + Bevacizumab | Capecitabine + Bevacizumab
Number analyzed (Participants) | 77 | 76
months | 18.0 [15.18 to 19.48] | 16.2 [13.07 to 17.67]
Statistical Analysis 1: Comparison: Trifluridine/Tipiracil + Bevacizumab vs Capecitabine + Bevacizumab; Test type: Other; p = 0.04, Cox proportional hazard model; Hazard Ratio (HR) = 0.56, 95% CI 2-sided [0.32 to 0.98]

ADVERSE EVENTS:
Time Frame: All Adverse Events (AE) were collected from the informed consent signature up to the final visit regardless of seriousness or relationship to study drug (maximum exposure: 82 weeks).
Description: Reported AEs are Treatment-Emergent AEs (TEAE) that are AEs that developed/worsened during the treatment period i.e. between the first treatment intake date and the last treatment intake date + 35 days.
  In the Capecitabine + bevacizumab group, the number of participants at Risk for TEAE (both serious and non-serious) was 76 which is different from Started patients in the Participant Flow module (=77). Indeed, 1 started patient in this group did not received any treatment dose
Arm/Group | Trifluridine/Tipiracil + Bevacizumab | Capecitabine + Bevacizumab
All-Cause Mortality (participants affected / at risk) | 22/77 | 33/76
Serious Adverse Events (participants affected / at risk) | 42/77 | 44/76
Other Adverse Events (participants affected / at risk) | 75/77 | 69/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trifluridine/Tipiracil + Bevacizumab (N=77) | Capecitabine + Bevacizumab (N=76)
Anaemia (Blood and lymphatic system disorders) | 3 (4) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3) | 3 (3)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 4 (5) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 5 (5)
Enterocutaneous fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal angiodysplasia haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Malignant bowel obstruction (Gastrointestinal disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (4) | 1 (1)
Death (General disorders) | 0 (0) | 2 (2)
General physical health deterioration (General disorders) | 0 (0) | 2 (2)
Mucosal dryness (General disorders) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatotoxicity (Hepatobiliary disorders) | 1 (1) | 0 (0)
Abdominal abscess (Infections and infestations) | 1 (1) | 0 (0)
Arthritis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Biliary sepsis (Infections and infestations) | 0 (0) | 1 (1)
Catheter site infection (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 2 (2) | 0 (0)
Device related sepsis (Infections and infestations) | 2 (2) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 2 (2) | 0 (0)
Peritonitis (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 1 (1)
Pneumonia toxoplasmal (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 2 (2)
Blood calcium decreased (Investigations) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1)
Blood magnesium decreased (Investigations) | 0 (0) | 1 (1)
Blood phosphorus decreased (Investigations) | 0 (0) | 1 (1)
Blood potassium decreased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1)
Troponin T increased (Investigations) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 5 (5)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (8) | 16 (16)
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1)
Cauda equina syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (3) | 2 (2)
Depressed mood (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (3) | 2 (2)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Female genital tract fistula (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (4)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 4 (4)
Hypertension (Vascular disorders) | 3 (3) | 0 (0)
Hypotension (Vascular disorders) | 1 (2) | 2 (2)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trifluridine/Tipiracil + Bevacizumab (N=77) | Capecitabine + Bevacizumab (N=76)
Anaemia (Blood and lymphatic system disorders) | 22 (31) | 5 (7)
Anaemia of chronic disease (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Anaemia of malignant disease (Blood and lymphatic system disorders) | 5 (5) | 1 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Haemolytic anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 6 (9) | 2 (5)
Neutropenia (Blood and lymphatic system disorders) | 40 (181) | 5 (5)
Spontaneous haematoma (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 11 (22) | 4 (5)
Thrombocytosis (Blood and lymphatic system disorders) | 4 (8) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Aortic valve thickening (Cardiac disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Bundle branch block right (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Dry eye (Eye disorders) | 1 (2) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 1 (1)
Eye pruritus (Eye disorders) | 0 (0) | 1 (1)
Lacrimation increased (Eye disorders) | 0 (0) | 4 (5)
Vision blurred (Eye disorders) | 1 (1) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 9 (18) | 6 (7)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (3) | 2 (3)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal inflammation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Aphthous ulcer (Gastrointestinal disorders) | 2 (2) | 1 (1)
Chronic gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 13 (21) | 15 (17)
Diarrhoea (Gastrointestinal disorders) | 40 (91) | 31 (64)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 6 (7)
Dyschezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 6 (7) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Eructation (Gastrointestinal disorders) | 2 (3) | 1 (1)
Gastrointestinal motility disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gingival bleeding (Gastrointestinal disorders) | 3 (4) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lip dry (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lip pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lip swelling (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mesenteric vein thrombosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 36 (84) | 13 (23)
Oral mucosa erosion (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis chronic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Periodontal disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 3 (6) | 3 (3)
Proctitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal discharge (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 13 (18) | 16 (29)
Stomatitis haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 22 (44) | 8 (8)
Asthenia (General disorders) | 14 (19) | 17 (22)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 3 (3)
Discomfort (General disorders) | 1 (1) | 0 (0)
Early satiety (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 28 (45) | 23 (35)
Feeling hot (General disorders) | 1 (1) | 0 (0)
Impaired healing (General disorders) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 3 (3) | 3 (3)
Injection site haematoma (General disorders) | 0 (0) | 1 (1)
Local swelling (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 1 (2) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 3 (4) | 3 (3)
Pain (General disorders) | 0 (0) | 1 (1)
Puncture site pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 5 (5) | 4 (5)
Tenderness (General disorders) | 0 (0) | 1 (1)
Xerosis (General disorders) | 0 (0) | 1 (1)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatomegaly (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 5 (7)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (2) | 3 (3)
Cystitis (Infections and infestations) | 0 (0) | 2 (2)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1)
Furuncle (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0)
Gastrointestinal viral infection (Infections and infestations) | 1 (1) | 0 (0)
Gingivitis (Infections and infestations) | 1 (1) | 0 (0)
Hepatic cyst infection (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 1 (1)
Labyrinthitis (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 1 (2) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1) | 3 (4)
Oral fungal infection (Infections and infestations) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 1 (1) | 4 (4)
Oral infection (Infections and infestations) | 1 (1) | 0 (0)
Periumbilical abscess (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 1 (1)
Rhinitis (Infections and infestations) | 4 (4) | 1 (1)
Skin candida (Infections and infestations) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 7 (8) | 2 (2)
Urinary tract infection (Infections and infestations) | 7 (8) | 5 (6)
Urinary tract infection bacterial (Infections and infestations) | 1 (1) | 2 (3)
Viral upper respiratory tract infection (Infections and infestations) | 8 (9) | 5 (5)
Vulvovaginal candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Abdominal wall wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 2 (5)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 5 (5) | 4 (6)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Stoma site irritation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Stoma site pain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 9 (11) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 7 (8) | 2 (2)
Bilirubin conjugated increased (Investigations) | 1 (2) | 1 (1)
Blood albumin decreased (Investigations) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 3 (3) | 2 (2)
Blood bilirubin increased (Investigations) | 6 (18) | 8 (13)
Blood bilirubin unconjugated increased (Investigations) | 0 (0) | 1 (1)
Blood cholesterol increased (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 3 (5) | 1 (1)
Blood glucose increased (Investigations) | 1 (1) | 0 (0)
Blood lactate dehydrogenase decreased (Investigations) | 1 (1) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 1 (5) | 4 (5)
Blood phosphorus increased (Investigations) | 1 (1) | 0 (0)
Blood potassium decreased (Investigations) | 0 (0) | 1 (1)
Blood potassium increased (Investigations) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 2 (3) | 0 (0)
Blood urea increased (Investigations) | 0 (0) | 1 (1)
Blood urine present (Investigations) | 0 (0) | 1 (1)
Carcinoembryonic antigen increased (Investigations) | 0 (0) | 1 (1)
Creatinine renal clearance decreased (Investigations) | 1 (1) | 1 (1)
Eosinophil count decreased (Investigations) | 2 (2) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 6 (6) | 2 (3)
Glomerular filtration rate decreased (Investigations) | 1 (1) | 0 (0)
Heart rate irregular (Investigations) | 0 (0) | 1 (1)
International normalised ratio increased (Investigations) | 1 (1) | 2 (2)
Lymphocyte count decreased (Investigations) | 4 (7) | 1 (2)
Monocyte count decreased (Investigations) | 2 (2) | 0 (0)
Neutrophil count decreased (Investigations) | 18 (90) | 1 (1)
Neutrophil count increased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 7 (22) | 3 (5)
Platelet count increased (Investigations) | 2 (3) | 0 (0)
Weight decreased (Investigations) | 9 (12) | 6 (7)
Weight increased (Investigations) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 15 (37) | 1 (1)
White blood cell count increased (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 29 (46) | 15 (23)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (6) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 4 (5) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 (4) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (4) | 1 (1)
Hypochloraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (8) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 7 (7)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 4 (5)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 (9) | 3 (3)
Amnesia (Nervous system disorders) | 0 (0) | 1 (1)
Aphonia (Nervous system disorders) | 0 (0) | 2 (2)
Balance disorder (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 5 (7) | 8 (10)
Dizziness exertional (Nervous system disorders) | 1 (1) | 1 (1)
Dizziness postural (Nervous system disorders) | 1 (1) | 1 (1)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 7 (8) | 8 (8)
Essential tremor (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 7 (13) | 4 (4)
Hyperaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (2)
Memory impairment (Nervous system disorders) | 1 (1) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (2) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 3 (3)
Neurotoxicity (Nervous system disorders) | 0 (0) | 1 (1)
Orthostatic intolerance (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 2 (3)
Restless legs syndrome (Nervous system disorders) | 1 (1) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2)
Confusional state (Psychiatric disorders) | 1 (1) | 1 (2)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Disorientation (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 6 (6) | 1 (1)
Mood altered (Psychiatric disorders) | 1 (1) | 0 (0)
Restlessness (Psychiatric disorders) | 1 (1) | 0 (0)
Stress (Psychiatric disorders) | 1 (1) | 0 (0)
Anuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 3 (3)
Glycosuria (Renal and urinary disorders) | 0 (0) | 1 (2)
Haematuria (Renal and urinary disorders) | 1 (1) | 2 (2)
Lower urinary tract symptoms (Renal and urinary disorders) | 1 (1) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 1 (1)
Nocturia (Renal and urinary disorders) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 5 (6) | 4 (5)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Oedema genital (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Catarrh (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (6)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 8 (11)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 4 (6)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 17 (17) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (4) | 4 (4)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Onychalgia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 3 (4) | 39 (49)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Skin fissures (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 9 (10) | 10 (12)
Hypotension (Vascular disorders) | 4 (5) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-01-25): https://cdn.clinicaltrials.gov/large-docs/21/NCT02743221/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-21): https://cdn.clinicaltrials.gov/large-docs/21/NCT02743221/SAP_001.pdf